CLINICAL TRIAL: NCT05361980
Title: Global Pediatric Orthopaedic Implant Safety & Efficacy Clinical Follow-up Program
Brief Title: Pediatric Orthopaedic Implant Safety & Efficacy
Acronym: Global POISE
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: OrthoPediatrics (Industry)
Responsible Party: Principal Investigator, Kishore Mulpuri, Professor, University of British Columbia
Other Study IDs: H21-03076
Record Dates: First submitted 2021-12-17; First posted 2022-05-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Fracture; Lengthening; Leg; Orthopedic Disorder; Deformity of Limb; Deformity; Bone; Implant Breakage; Implant Complication; Hip Dysplasia; Pediatric ALL; Hip Disease; Hip Dislocation
MeSH Terms: conditions — Fractures, Bone; Musculoskeletal Diseases; Congenital Abnormalities; Hip Dislocation; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Longitudinal Observational Group: Pediatric patients indicated for the device-specific indication, per physician discretion and as indicated in the device IFU.
  Interventions: Device: Pediatric orthopaedic implant

INTERVENTIONS:
Device: Pediatric orthopaedic implant — Patient receives a pediatric orthopaedic implant as a part of standard clinical care.

SUMMARY:
Implant devices are important tools - their use is essential across a number of orthopaedic indications, including hip conditions, trauma and limb deformity.

Given the vital role fixation devices play in maintaining alignment, promoting healthy bone healing and preventing joint degeneration, it is essential to understand the expected lifetime outcomes of these implants, and evaluate their safety and efficacy.

Prospective implant efficacy and safety registries are needed to support this endeavour, especially considering new regulatory requirements from the European Union Medical Devices Regulation (EU MDR) in relation to post-market clinical follow-up (PMCF).

DETAILED DESCRIPTION:
STUDY PROCEDURES Screening Patients will be screened against basic inclusion/exclusion criteria to see if patients may be appropriate for study participation according to any standard of care assessments available, and where appropriate with the site's REB/IRB screening procedures and local regulatory requirements. If a patient is deemed eligible, data outlined throughout this protocol will be collected, de-identified and entered into a Research Electronic Database Capture (REDCap) system managed at BCCH.

Enrollment Patients will be assigned a sequential, unique study number (subject ID) and de-identified data will be entered in the study database. The center number is designated by the BCCH team for each individual investigational site. The patient number will be in sequential order by the patient screening date starting with 001. Once a patient has been assigned a subject ID, the number will not be reused.

Pre-Operative Procedures Once a patient is identified as eligible for an Implant Safety and Efficacy device report, it will be determined whether that patient is already enrolled in one of the existing condition-specific registries. Should participants be enrolled in a condition-specific registry, demographic data, medical history, preoperative clinical data, including any pre-existing infections at or near the operative site, and data on pre-operative radiographs for the relevant underlying diagnosis will have already been prospectively collected under registry procedures. If a patient has not been previously enrolled in a condition-specific registry, the patient will be offered enrollment in both the condition registry and for the purposes of the Implant Safety and Efficacy device report. Demographic data, medical history, preoperative clinical data and data on pre-operative radiographs for the relevant underlying diagnosis will then be collected retrospectively from the medical record.

Required Data Collection:

Operative details in the source documentation will be collected that provide specific information from the subject's surgery such as surgical approach, complications, and unique device identification (UDI) numbers for the implanted device.

The following data will be collected and entered into the registry:

* Operative data, specific to the technique related to the relevant OrthoPediatrics system/device
* Assessments of any device-related adverse events
* Assessment for other adverse events
* When possible, the UDI number for the device(s) implanted, or information on the device implanted

Follow-up Procedures

Data collected during routine standard of care follow-up visits will be collected as part of this study. The following data will be collected:

* Radiographs obtained during study clinical evaluations to determine bony union, as well as healing or complications
* Device-related adverse events
* Unanticipated device-related serious adverse device effects
* Information on implant removals not related to an adverse event; degree of bony union just prior to implant removal Unscheduled Visits [if or when needed]

The condition-specific registries are designed to capture every visit that occurs, whether scheduled or unscheduled. An unscheduled visit may occur when an adverse event occurs, or when a patient returns outside of the planned interval window. If an unscheduled visit occurs, the following assessments are to be done:

* Assessment of any adverse events related to the device
* Survivorship of the device

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for the device-specific indication, per physician discretion and as indicated in the device IFU. Off-label use is strongly discouraged; however, any and all on- and off-label indications for use of the products in this program will be collected and stratified accordingly
* Patients must be able to adhere to the required length of follow-up for the endpoints of each individual product
* Informed consent/assent is required

Exclusion Criteria:

* Patients with a demonstrated sensitivity to metals
* Patients with an inability to follow a post-operative regimen

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Anyone who meets the eligibility criteria and is within the age limits listed in the above sections can participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Device related adverse events | 2 years post implant insertion
  Determine the frequency and severity of device-related adverse events at device-specific end points. All adverse events will be recorded and followed during the study. The frequency and severity of device related adverse events will be analyzed to ensure the device risk profile has not changed.
Implant survival | 2 years post implant insertion
  Determine the implant survival rate at post-operative end-point: (lack of revision)
Implant efficacy | 2 years post implant insertion
  Efficacy will be assessed by post-operative clinical and radiographic evaluations at each follow-up end-point to assess bone fixation and/or deformity correction.

SECONDARY OUTCOMES:
Numeric pain rating scale (NPRS) | 2 years post implant insertion
  The numeric pain rating scale (NPRS) is a subjective, 11-point numerical scale in which respondents self-report their pain on a scale of 0 (no pain at all) to 10 (worst pain imaginable).
LIMB-Q Kids | 2 years post implant insertion
  LIMB-Q Kids is a new patient reported outcome measure (PROM) for children with lower limb deformities.
PROMIS | 2 years post implant insertion
  The Patient Reported Outcomes Measurement Information System (PROMIS) measures are self-reported and parent-reported. It includes over 300 measures of global, physical, mental, and social health for adults and children in the general population and those living with a chronic condition. Specifically, the PROMIS Global Health will be administered to all patients while the PROMIS Physical Function - Mobility short form will be administered to those with an implant used in a lower extremity and the PROMIS Physical Function - Upper Extremity short form will be administered to those with an implant used in an upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Bryn Zomar, PhD, Study Director — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No